CLINICAL TRIAL: NCT01554371
Title: A Phase Ib/II Study of Eribulin in Combination With Cyclophosphamide in Patients With Solid Tumor Malignancies
Brief Title: Eribulin in Combination With Cyclophosphamide in Patients With Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11996; NCI-2012-00436 (Registry Identifier: Clinical Trials Reporting Program)
Record Dates: First submitted 2012-03-09; First posted 2012-03-15 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Malignant Solid Tumour; Breast Cancer Nos Metastatic Recurrent; Neuropathy
Keywords: Solid tumor; Metastatic breast cancer; Unresectable or metastatic carcinoma; Neuropathy; Eribulin; Cyclophosphamide
MeSH Terms: conditions — Breast Neoplasms; Carcinoma | interventions — eribulin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1b: 1.1 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) (Experimental): Dose escalation cohort will include all patients with solid tumors. Eribulin mesylate 1.1 mg/ m2 on days 1 and 8 followed by cyclophosphamide 600 mg/m2 on day 1 of a 21-day cycle.The highest dose level at which no more than one of six subjects experience DLT defines the MTD
  Interventions: Drug: Eribulin; Drug: Cyclophosphamide
- Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) (Experimental): Dose escalation cohort will include all patients with solid tumors. Eribulin mesylate 1.4 mg/ m2 on days 1 and 8 followed by cyclophosphamide 600 mg/ m2 on day 1 of a 21-day cycle.The highest dose level at which no more than one of six subjects experience DLT defines the MTD
  Interventions: Drug: Eribulin; Drug: Cyclophosphamide
- Phase II: Eribulin Combination w/ Cyclophosphamide (Breast Cancer Expansion Cohort) (Experimental): Dose-expansion cohort will enroll patients with advanced breast cancer only after Phase Ib enrollment has been concluded. The MTD of Eribulin mesylate will be administered on days 1 and 8 followed by cyclophosphamide 600 mg/m2 on day 1 of a 21-day cycle.
  Interventions: Drug: Eribulin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Eribulin — Given intravenously (IV)
  Phase II: Eribulin mesylate (mg/m2) + Cyclophosphamide (mg/ m2) for advanced breast cancer participants only
  Other Names: Halaven; E7389; ER-086526
Drug: Cyclophosphamide — Given IV
  Other Names: Cytoxan

SUMMARY:
The purpose of this study is to test the safety of eribulin (Halaven™) and cyclophosphamide (Cytoxan®) given together at different doses. This study will look at what effects, good and/or bad, that these drugs have on solid tumors. Eribulin is a drug that has been approved by the FDA for breast cancer that has spread to other parts of the body. Cyclophosphamide has been approved for different types of cancers (including breast cancer). However, the combination of eribulin and cyclophosphamide is considered experimental; that means this combination has not been approved by the FDA.

The funding for this study is provided by Eisai Inc., the maker of eribulin.

DETAILED DESCRIPTION:
This is a phase Ib/II trial designed to determine the maximum tolerated dose (MTD) and does limiting toxicities (DLTs) of the combination of eribulin and cyclophosphamide in solid tumors and make preliminary estimates regarding efficacy of this treatment in patients with advanced breast cancer.

The study includes a standard dose-confirmation schema (phase Ib portion) enrolling 3 to 6 patients/subjects, with any solid tumors, per cohort (3+3 design) with a total of 18 patients. The dose-expansion (phase II portion) will enroll 40 patients with advanced breast cancer to detect an effect size of 15% with a power of 80% with endpoints of safety, efficacy, and clinical benefit rate. A maximum of 58 patients will be enrolled on the phase Ib and II portions of this trial combined and will be treated until disease progression or toxicity mandate treatment change.

Eribulin is a non-taxane microtubule inhibitor that is FDA approved as monotherapy for the treatment of taxane and anthracycline resistant metastatic breast cancer. The combination of docetaxel and cyclophosphamide is a well-accepted adjuvant chemotherapy regimen that has become an increasingly common therapeutic choice for intermediate risk early stage breast cancer. Eribulin has a favorable toxicity profile compared to docetaxel with the most common adverse reactions (incidence ≤25%) including neutropenia, anemia, asthenia/fatigue, alopecia, peripheral neuropathy, nausea, and constipation. Eribulin appears to have activity in taxane resistant disease, making it an attractive partner with cyclophosphamide.

Neuropathy can be a devastating complication from adjuvant chemotherapy and in the metastatic setting, may limit effective therapy and reduce quality of life. Understanding the host factors that predict risk for neuropathy is critical, as these patients may in particular benefit from the lower risk of neuropathy associated with eribulin therapy. In conjunction with this trial, we have included correlative studies to study the proposed pharmacogenomic factors associated with risk of neuropathy. In this way we will potentially be able to identify patients who could preferentially be treated with less neurotoxic microtubule inhibitors.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Phase Ib: Patient must have histologically or cytologically documented solid tumor malignancies.

   Phase II: Patients must have histologically or cytologically confirmed locally advanced, unresectable or metastatic carcinoma of the breast.
2. Patient is male or female and ≥18 years of age on the day of signing informed consent.
3. Patient must have performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale and life expectancy > 3 months.
4. Patient must have evaluable disease. Measureable disease is not required
5. Patient must have adequate organ function
6. Female patient of childbearing potential must have a negative serum or urine pregnancy test quantitative human chorionic gonadotropin (β-hCG) within 72 hours prior to receiving the first dose of study medication and agree to the use of effective methods of contraception while on study.
7. Any number of prior lines of chemotherapy in the metastatic setting is allowed.
8. Concomitant use of bisphosphonates is allowed.
9. Patients with stable and clinically insignificant CNS disease are allowed. Patients must be off steroids with no new CNS symptoms or findings on radiographic imaging for 1 month.
10. Patients willing and able to complete the questionnaires.
11. Patients willing and able to comply with the study protocol for the duration of the study.
12. Written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

EXCLUSION CRITERIA:

1. Patients who have had chemotherapy or radiotherapy within two weeks, 4 weeks for nitrosoureas, mitomycin C, pegylated-doxorubicin and one half-life for bevacizumab, hormone therapy within one week, trastuzumab within 2 weeks or lapatinib within one week of study Day 1.
2. If the patient has residual toxicity from prior treatment, toxicity must be ≤ Grade 1.
3. Patients with non-healing surgical wounds. Patients must be at least two weeks from a major surgical procedure, and surgical wounds must be completely healed.
4. Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis. However, patients with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for at least 1 month prior to entry as defined as:

   1. no evidence of new or enlarging CNS metastasis
   2. off steroids that are used to minimize surrounding brain edema. Patients with clinically insignificant brain metastases that do not require treatment are eligible.
5. Patients with known hypersensitivity to the components of study drug or its analogs.
6. Significant cardiovascular impairment:

   1. Congestive heart failure, Clinically significant cardiac arrhythmia, history or current evidence of a myocardial infarction during the last 6 months, and/or a current ECG tracing that is abnormal in the opinion of the treating Investigator, or unstable angina
   2. QTc prolongation >480 msec (Bazett's Formula) or congenitally long QT syndrome (LQTS)
7. Severe/uncontrolled concurrent illness/infection
8. Patients with other active, current primary malignancies, other than carcinoma in situ of the cervix or non-melanoma skin cancer
9. Patients with > Grade 1 neuropathy at screening
10. Patients with a hypersensitivity to halichondrin B and/or halichondrin B chemical derivative
11. Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
12. Patients with other significant disease or disorders that, in the Investigator's opinion, would exclude the patient from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-03-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S Rugo, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gumusay O, Huppert LA, Magbanua MJM, Wabl CA, Assefa M, Chien AJ, Melisko ME, Majure MC, Moasser M, Park J, Rugo HS. A phase Ib/II study of eribulin in combination with cyclophosphamide in patients with advanced breast cancer. Breast Cancer Res Treat. 2024 Jan;203(2):197-204. doi: 10.1007/s10549-023-07073-0. Epub 2023 Oct 10. PMID 37815684

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b: 1.1 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort): Dose escalation cohort will include all patients with solid tumors. Eribulin mesylate 1.1 mg/ m2 on days 1 and 8 followed by cyclophosphamide 600 mg/ m2 on day 1 of a 21-day cycle.The highest dose level at which no more than one of six subjects experience DLT defines the MTD
  Eribulin: Given intravenously (IV) Cyclophosphamide: Given IV
- Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort): Dose escalation cohort will include all patients with solid tumors. Eribulin mesylate 1.4 mg/ m2 on days 1 and 8 followed by cyclophosphamide 600 mg/ m2 on day 1 of a 21-day cycle.The highest dose level at which no more than one of six subjects experience DLT defines the MTD
  Eribulin: Given intravenously (IV) Cyclophosphamide: Given IV
- Phase II: Eribulin Combination w/ Cyclophosphamide (Breast Cancer Expansion Cohort): Dose-expansion cohort will enroll patients with advanced breast cancer only after Phase Ib enrollment has been concluded. The MTD of Eribulin mesylate will be administered on days 1 and 8 followed by cyclophosphamide 600 mg/m2 on day 1 of a 21-day cycle.
  Eribulin: Given intravenously (IV) Cyclophosphamide: Given IV
Period: Overall Study
Arm/Group | Phase 1b: 1.1 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) | Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) | Phase II: Eribulin Combination w/ Cyclophosphamide (Breast Cancer Expansion Cohort)
Started | 3 | 3 | 38
Completed | 3 | 3 | 38
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b: 1.1 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort): Dose escalation cohort will include all patients with solid tumors. Eribulin mesylate 1.1 mg/m2 on days 1 and 8 followed by cyclophosphamide 600 mg/m2 on day 1 of a 21-day cycle. The highest dose level at which no more than one of six subjects experience DLT defines the MTD
  Eribulin: Given intravenously (IV) Cyclophosphamide: Given IV
- Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort): Dose escalation cohort will include all patients with solid tumors. Eribulin mesylate 1.4 mg/m2 on days 1 and 8 followed by cyclophosphamide 600 mg/m2 on day 1 of a 21-day cycle. The highest dose level at which no more than one of six subjects experience DLT defines the MTD
  Eribulin: Given intravenously (IV) Cyclophosphamide: Given IV
- Total: Total of all reporting groups
Arm/Group | Phase 1b: 1.1 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) | Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) | Phase II: Eribulin Combination w/ Cyclophosphamide (Breast Cancer Expansion Cohort) | Total
Number analyzed (Participants) | 3 | 3 | 38 | 44
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 0 | 0 | 1 | 1
  40-49 years old | 1 | 2 | 12 | 15
  50-59 years old | 1 | 0 | 10 | 11
  60-69 years old | 1 | 1 | 11 | 13
  70-79 years old | 0 | 0 | 3 | 3
  80-89 years old | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 38 | 44
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 2 | 3 | 36 | 41
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 3
  White | 3 | 2 | 29 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 38 | 44

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) in Participants With Any Solid Tumor (Phase Ib)
Description: Standard dose-confirmation design of 3 to 6 participants per cohort (3+3 design) was used to determine the MTD of eribulin in combination with cyclophosphamide for participants with any solid tumor. The highest dose level or MTD is reached when no more than one of six participants experience a Dose Limiting Toxicity (DLTs). A DLT is defined as any treatment-related toxicity in first 28 days of therapy with a grade 3 or 4 non-hematologic toxicity, a grade 4 neutropenia or thrombocytopenia lasting >7 days or febrile neutropenia, or any clinically significant toxicity grade 2 or higher that requires more than 14 days to resolve. The highest dose level at which no more than one of six participants experience DLT defines the MTD.
Time Frame: Up to 24 months
Measure: Number; unit: milligrams per square meter (mg/m2)
Groups:
- Phase 1b: Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort): Dose escalation cohort will include all patients with solid tumors. Eribulin mesylate 1.1 mg/ m2 on days 1 and 8 followed by cyclophosphamide 600 mg/ m2 on day 1 of a 21-day cycle.The highest dose level at which no more than one of six subjects experience DLT defines the MTD
  Eribulin: Given intravenously (IV) Cyclophosphamide: Given IV
Arm/Group | Phase 1b: Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort)
Number analyzed (Participants) | 6
milligrams per square meter (mg/m2)
  Eribulin | 1.4
  Cyclophosphamide | 600

2. Primary Outcome: Clinical Benefit Rate for Patients With Advanced Breast Cancer (ABC) (Phase II)
Description: The clinical benefit rate is defined as the proportion of participants with confirmed complete response (CR), partial response (PR) and stable disease (SD) evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Responses are determined by changes in the largest diameter of the tumor lesions and the shortest diameter in the case of malignant lymph nodes. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter, PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters, and SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Only participants with measurable disease present at baseline, received at least 1 cycle of therapy, and had disease re-evaluated will be considered evaluable.
Time Frame: Up to 24 months
Measure: Number; unit: proportion of particpants
Arm/Group | Phase II: Eribulin Combination w/ Cyclophosphamide (Breast Cancer Expansion Cohort)
Number analyzed (Participants) | 38
proportion of particpants | .135

3. Secondary Outcome: Number of Participants With Treatment-related Toxicities
Description: Safety of combination of eribulin and cyclophosphamide in participants was assessed by monitoring the frequency of treatment-related toxicities according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 with an attribute of possibly, probably, or definitely related to treatment. Number of participants by toxicity will be reported.
Time Frame: Up to 24 months
Measure: Number; unit: participants
Groups:
- Phase 1b: 1.1 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort): Dose escalation cohort will include all patients with solid tumors. Eribulin mesylate 1.1 mg/ m2 on days 1 and 8 followed by cyclophosphamide 600 mg/m2 on day 1 of a 21-day cycle.The highest dose level at which no more than one of six subjects experience DLT defines the MTD
  Eribulin: Given intravenously (IV) Cyclophosphamide: Given IV
- Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort): Dose escalation cohort will include all patients with solid tumors. Eribulin mesylate 1.4 mg/ m2 on days 1 and 8 followed by cyclophosphamide 600 mg/m2 on day 1 of a 21-day cycle.The highest dose level at which no more than one of six subjects experience DLT defines the MTD
  Eribulin: Given intravenously (IV) Cyclophosphamide: Given IV
Arm/Group | Phase 1b: 1.1 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) | Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) | Phase II: Eribulin Combination w/ Cyclophosphamide (Breast Cancer Expansion Cohort)
Number analyzed (Participants) | 3 | 3 | 38
participants
  Nausea | 3 | 3 | 19
  Constipation | 3 | 1 | 0
  Fatigue | 1 | 3 | 26
  Peripheral sensory neuropathy | 2 | 1 | 15
  Anorexia | 1 | 2 | 13
  White blood cell decreased | 1 | 2 | 18
  Mucositis oral | 1 | 1 | 3
  Platelet count decreased | 0 | 2 | 5
  Alopecia | 1 | 1 | 9
  Arthralgia | 1 | 1 | 2
  Hemoglobin increased | 0 | 1 | 0
  Headache | 1 | 0 | 4
  Chills | 0 | 1 | 3
  Alanine aminotransferase increased | 1 | 0 | 0
  Rash maculo-papular | 0 | 1 | 3
  Epistaxis | 1 | 0 | 0
  Hypomagnesemia | 1 | 0 | 3
  Edema limbs | 1 | 0 | 3
  Vomiting | 1 | 0 | 10
  Abdominal pain | 0 | 1 | 3
  Anemia | 0 | 0 | 13
  Investigations - Other | 0 | 1 | 5
  Dysgeusia | 1 | 0 | 0
  Alkaline phosphatase increased | 1 | 0 | 2
  Hoarseness | 1 | 0 | 2
  Fever | 0 | 1 | 8
  Neutrophil count decreased | 0 | 0 | 23
  Diarrhea | 0 | 0 | 10
  Hypokalemia | 0 | 0 | 8
  Weight loss | 0 | 0 | 8
  Gastrointestinal disorders - Other | 0 | 0 | 6
  Nasal congestion | 0 | 0 | 5
  Cough | 0 | 0 | 5
  Upper respiratory infection | 0 | 0 | 5
  Sinusitis | 0 | 0 | 3
  Febrile neutropenia | 0 | 0 | 3
  Bone pain | 0 | 0 | 3
  Blurred vision | 0 | 0 | 3
  Peripheral motor neuropathy | 0 | 0 | 3
  Dyspnea | 0 | 0 | 3
  Gastroesophageal reflux disease | 0 | 0 | 3
  Lymphocyte count decreased | 0 | 0 | 2
  Dizziness | 0 | 0 | 2
  Hypoalbuminemia | 0 | 0 | 2
  Hot flashes | 0 | 0 | 2
  Aspartate aminotransferase increased | 0 | 0 | 2
  Memory impairment | 0 | 0 | 2
  Postnasal Drip | 0 | 0 | 2
  Insomnia | 0 | 0 | 2
  Pain | 0 | 0 | 2
  Non-cardiac chest pain | 0 | 0 | 2
  Hypoxia | 0 | 0 | 1
  Portal vein thrombosis | 0 | 0 | 1
  Sepsis | 0 | 0 | 1
  Confusion | 0 | 0 | 1
  Hypophosphatemia | 0 | 0 | 1
  Pain in extremity | 0 | 0 | 2
  Hypercalcemia | 0 | 0 | 1
  Dysphagia | 0 | 0 | 1
  Hyponatremia | 0 | 0 | 1
  Myalgia | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) for Participants With Any Solid Tumor (Phase 1b)
Description: For the purposes of Phase Ib dose escalation, DLTs will be defined as any treatment-related toxicity occurring within the first 21 days of combination therapy as grade 3 or 4 clinically evident non-hematologic toxicity; grade 4 neutropenia or thrombocytopenia lasting > 7 days or febrile neutropenia; or any clinically significant toxicity grade 2 or higher that requires more than 14 days to resolve.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid: Dose escalation cohort will include all patients with solid tumors. Eribulin mesylate 1.4 mg/ m2 on days 1 and 8 followed by cyclophosphamide 600 mg/m2 on day 1 of a 21-day cycle.The highest dose level at which no more than one of six subjects experience DLT defines the MTD
  Eribulin: Given intravenously (IV) Cyclophosphamide: Given IV
Arm/Group | Phase 1b: 1.1 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) | Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

5. Secondary Outcome: Overall Response Rate (ORR) for Participants With Advanced Breast Cancer (Phase II)
Description: The ORR is defined as the proportion of participants displaying a CR or PR per RECIST criteria recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The participant's best response will depend on the achievement of both measurement and confirmation criteria with CR defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter and PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 24 months
Measure: Number; unit: proportion of participants
Arm/Group | Phase II: Eribulin Combination w/ Cyclophosphamide (Breast Cancer Expansion Cohort)
Number analyzed (Participants) | 38
proportion of participants | .131

6. Secondary Outcome: Time to Progression for Participants With Advanced Breast Cancer (Phase II)
Description: Time to progression will be evaluated as time from first treatment to tumor progression in weeks. Disease progression will be measured using Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (uni-dimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST 1.1 criteria.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase II: Eribulin Combination w/ Cyclophosphamide (Breast Cancer Expansion Cohort)
Number analyzed (Participants) | 38
weeks | 16.4 [13.8 to 21.1]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Phase 1b: 1.1 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) | Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) | Phase II: Eribulin Combination w/ Cyclophosphamide (Breast Cancer Expansion Cohort)
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/3 | 32/38
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 5/38
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: 1.1 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) (N=3) | Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) (N=3) | Phase II: Eribulin Combination w/ Cyclophosphamide (Breast Cancer Expansion Cohort) (N=38)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Low Hematocrit (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: 1.1 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) (N=3) | Phase 1b: 1.4 mg/m2 Eribulin Combination w/ Cyclophosphamide (Solid Tumor Escalation Cohort) (N=3) | Phase II: Eribulin Combination w/ Cyclophosphamide (Breast Cancer Expansion Cohort) (N=38)
Nausea (Gastrointestinal disorders) | 3 (5) | 3 (6) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 8 (10)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 4 (7)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (4) | 0 (0)
Edema Limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 7 (9)
Pain (General disorders) | 0 (0) | 0 (0) | 7 (12)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (7) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 2 (6) | 0 (0)
Investigations - Other (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight Loss (Investigations) | 0 (0) | 0 (0) | 10 (12)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (5)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (6)
Hemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 12 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 11 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 8 (10)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 18 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 9 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 9 (10)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (7)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 9 (20)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 11 (12)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 9 (9)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 6 (6)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 6 (6)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 3 (5)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 2 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT01554371/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT01554371/ICF_001.pdf